CLINICAL TRIAL: NCT01242059
Title: Effect of Yellow Pea Fractions on Short-term Food Intake at 120 Minutes, Subjective Appetite and Glycemic Response in Young Adult Males
Brief Title: Yellow Pea Fractions and Short-term Food Intake, Subjective Appetite and Glycemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government); Pulse Canada (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: PureNet_23281
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Obesity; Type II Diabetes Mellitus; Metabolic Syndrome
Keywords: Obesity; Food intake regulation; blood glucose regulation; protein; fiber; pulses; yellow peas
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control Tomato Soup (Experimental)
  Interventions: Dietary Supplement: Control
- 10 g of yellow pea fiber (Experimental)
  Interventions: Other: yellow pea fiber
- 20 g of yellow pea fiber (Experimental)
  Interventions: Other: yellow pea fiber
- 10 g of yellow pea protein (Experimental)
  Interventions: Dietary Supplement: yellow pea protein
- 20 g of yellow pea protein (Experimental)
  Interventions: Dietary Supplement: yellow pea protein

INTERVENTIONS:
Dietary Supplement: yellow pea protein — Served in a tomato soup
  Arms: 10 g of yellow pea protein; 20 g of yellow pea protein
Other: yellow pea fiber — Served in a tomato soup
  Arms: 10 g of yellow pea fiber; 20 g of yellow pea fiber
Dietary Supplement: Control — Served in a tomato soup
  Arms: Control Tomato Soup

SUMMARY:
It is hypothesized that yellow pea protein and fiber will reduce short-term food intake, subjective appetite and glycemic response.

DETAILED DESCRIPTION:
A within-subject, randomized study was conducted. Each subject returned 5 times, 1 week apart, and received 1 of the 5 treatments per week. The 5 treatments were tomato soup with 10 or 20 g of isolated yellow pea fibre or protein, or a control soup with no added pea fractions. Food intake was measured at an ad libitum pizza meal served 2 hours after treatment. Satiety and blood glucose (via finger prick) were measured throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* male 20-30 years old healthy weight

Exclusion Criteria:

* smoking restrictive eating metabolic diseases breakfast skippers dieters

Ages: 20 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Energy Intake | at 120 minutes after treatment
  Energy intake at an ad libitum pizza meal

SECONDARY OUTCOMES:
Glycemic Response | 200 minutes
Subjective Appetite | 200 minutes

CONTACTS AND LOCATIONS:
Overall Officials: G Harvey Anderson, Ph.D, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto - Department of Nutritional Sciences, Toronto, Ontario, Canada